CLINICAL TRIAL: NCT00898287
Title: A Phase I/II Study to Evaluate Safety and Efficacy of P276-00 in Combination With Gemcitabine in Patients With Cancer of Pancreas
Brief Title: Safety and Efficacy Study of P276-00 in Combination With Gemcitabine in Patients With Advanced Pancreatic Cancer
Acronym: SAVIOR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/28/08; P276-00/28/08
Record Dates: First submitted 2009-05-06; First posted 2009-05-12 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Pancreatic Cancer
Keywords: Locally advanced or metastatic adenocarcinoma of pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — P276-00; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- P276-00 plus Gemcitabine (Experimental): Subjects will be enrolled at different levels of P276-00 dosage as follows:- Level 1 - 100mg/m2/day x 5 q 3 weeks Level 2 - 140 mg/m2/day x 5 q 3 weeks Level 3 - 185 mg/m2/day x 5 q 3 weeks P276-00 will be administered as intravenous infusion in 200 ml of 5% dextrose over 30min from days 1 to 5 per 21 day cycle. Six such cycles will be administered unless there is progression of disease or unacceptable toxicity.
  Gemcitabine will be administered as an intravenous infusion at dose of 1000mg/m2 over 30 mins every week for 7 weeks followed by a gap of one week and then 3 weekly doses every 4 weeks. This treatment will be continued for six P276-00 cycles of 3 weeks each unless there is progression of disease or unacceptable toxicity.
  Interventions: Drug: P276-00; Drug: Gemcitabine

INTERVENTIONS:
Drug: P276-00 — Subjects will be enrolled at different levels of P276-00 dosage as follows:- Level 1 - 100mg/ m 2/day x 5 q 3 weeks Level 2 - 140 mg/ m2/day x 5 q 3 weeks Level 3 - 185 mg/ m2 /day x 5 q 3 weeks P276-00 will be administered as intravenous infusion in 200 ml of 5% dextrose over 30min from days 1 to 5 per 21 day cycle. Six such cycles will be administered unless there is progression of disease or unacceptable toxicity.
Drug: Gemcitabine — Gemcitabine will be administered as an intravenous infusion at dose of 1000mg/m 2 over 30 mins every week for 7 weeks followed by a gap of one week and then 3 weekly doses every 4 weeks. This treatment will be continued for six P276-00 cycles of 3 weeks each unless there is progression of disease or unacceptable toxicity.

SUMMARY:
The purpose of this study is to identify a dose of P276-00 that can be safely administered along with Gemcitabine and to examine safety and efficacy of the combination in treatment of advanced pancreatic cancer.

DETAILED DESCRIPTION:
This study is an open label multicenter trial to evaluate safety and efficacy of P276-00 in combination with Gemcitabine in subjects with locally advanced or metastatic pancreatic cancer. Primary objective in part A is to determine maximum tolerated dose (MTD) of P276-00 in combination with Gemcitabine and in part B to evaluate efficacy of this combination in subjects with locally advanced or metastatic pancreatic cancer. In part A, cohort of 3 subjects will be enrolled at starting dose level of P276-00 which is 100 mg/m2/ day to be given intravenously (IV) from day 1 to day 5 every 21 days. This constitutes one cycle of P276-00. If this dose is well tolerated then next cohort will be enrolled at higher dose level of P276-00. P276-00 dose escalation will continue until MTD of P276-00 in combination with Gemcitabine is determined. The subsequent dose levels of P276-00 will be 140 mg/m2/day and 185 mg/m2/day. In part B ten subjects will be evaluated at the MTD of P276-00 in combination with Gemcitabine to evaluate efficacy of the combination. Dose of Gemcitabine will be same in both parts of the study which is 1000mg/m2 over 30mins every week for 7 weeks followed by a gap of one week and then 3 weekly doses every 4 weeks. Subjects will be treated for six cycles of P276-00 in combination with Gemcitabine or until evidence of disease progression or unacceptable toxicity. Safety evaluations will be performed at regular intervals by means of record of vital parameters, physical examination and laboratory investigations for hematology and biochemistry. Efficacy assessment will be performed by means of weekly record of pain intensity, analgesic consumption, change in weight and performance status for evaluation of clinical benefit response and by means of CT scans at the end of every 2 cycles for evaluation of tumor response by RECIST (Response Evaluation Criteria in Solid Tumors)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of infiltrating ductal adenocarcinoma of pancreas.
2. Chemonaive patients i.e. patients must not have received chemotherapy or biologic/targeted anticancer therapy for the adenocarcinoma of pancreas.
3. Locally advanced inoperable pancreatic cancer.
4. Patients of either sex, aged > or = 18 years.
5. Karnofsky performance status of > or = 60%.
6. Adequate bone marrow reserve: white blood cell (WBC) count > or = 4 x 109/l, Absolute neutrophil count (ANC) ≥ 1.5 x 109/l, platelets > or = 100 x 109/l, hemoglobin > or = 10 g/dl.
7. Adequate liver function: bilirubin < or = 1.5 times the upper normal value, ALT/AST/ alkaline phosphatase less than 3 times the upper normal value (unless due to liver metastases in which case bilirubin less than 3 times the upper normal value, ALT/AST less than 4 times the upper normal value, and alkaline phosphatase without limit).
8. Adequate renal function: creatinine ≤ 1.5 times the upper normal value.
9. If female:

   * Childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of at least 2 approved contraceptive methods (at least one should be a barrier method) during and for 4 weeks after stopping the study treatment.
   * Negative urine β-HCG test within 1 week prior to protocol entry where childbearing potential is not terminated.
10. Additional inclusion criterion only for part B: Patient should satisfy at least one of the following criteria on cycle 1 day 1:

    * Karnofsky performance status of 60 or 70
    * Baseline pain intensity score of > or = 20 mm

Exclusion Criteria:

1. Inability / unwillingness to give consent.
2. Pregnant or breast feeding women.
3. Brain metastasis (active or inactive).
4. Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
5. Patients known to be suffering from infection with HIV, Hepatitis C or Hepatitis B.
6. Patients who had received any other investigational drug within 1 month prior to Day 1 of protocol treatment.
7. Patients with QTc > 450 msec on 12-lead standard electrocardiogram (ECG).
8. Major surgery within 2 weeks prior to protocol treatment.
9. Radiotherapy to > 10% of bone marrow.
10. Patients with 3rd space fluid accumulation (ascites, pleural effusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of P276-00 administered along with Gemcitabine. | 3 weeks

SECONDARY OUTCOMES:
To evaluate pharmacokinetic parameters of P276-00. | one week
To determine clinical benefit response to P276-00 in combination with Gemcitabine in patients with cancer of pancreas. | Every week
To determine objective tumor response rate to P276-00 in combination with Gemcitabine in patients with cancer of pancreas. | Every 6 weeks
To characterize toxicities of P276-00 in combination with Gemcitabine. | Every week

CONTACTS AND LOCATIONS:
Overall Officials: Amol Bapaye, MS, Principal Investigator — Deenanath Mangeshkar Hospital & Research Centre, ,Pune, India; Raj Nagarkar, MS, Principal Investigator — Curie Manavata Cancer Centre, Nashik, India; J S Rajkumar, DNB, Principal Investigator — Lifeline Mutispecilaity Hospital, Chennai, India; Ravi K Saxena, DNB, Principal Investigator — Global Hospital, Hyderabad, India.; Kirushna Kumar, MD, Principal Investigator — Meenakshi Mission Hospital & Reasearch Centre, Madurai, India; Anita Ramesh, MD, Principal Investigator — Sri RamaChandra Medical Centre, Chennai, India; Ajay Mehta, MS, Principal Investigator — Central India cancer Research Institute, Nagpur, India
Locations (7):
- India (7):
  - Central India Cancer Research Institute, Nagpur, Ajayonco@hotmail.com
  - Global Hospital, Hyderabaad, Andhra Pradesh
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Sri RamaChandra Medical Centre, Chennai, Tamil Nadu
  - Lifeline Mutispecilaity Hospital, Chennai, Tamil Nadu
  - Meenakshi Mission Hospital & Reasearch Centre, Madurai, Tamil Nadu